CLINICAL TRIAL: NCT02471001
Title: Coronary Sinus Blood Isoflurane Concentration in Patients Undergoing Heart Surgery
Brief Title: The Levels of Anaesthetics in Heart Muscle During Heart Surgery
Acronym: TLAHMHS
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: UEdin-15
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Surgery
Keywords: concentration; Isoflurane; cardioprotective; cardioplegia; heart surgery; Disorder; Heart; Functional; Postoperative
MeSH Terms: conditions — Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Surgery Using Heart-lung Machine: All patients who scheduled for an elective heart surgery in Royal Infirmary of Edinburgh using a heart-lung machine and the administration of ether-like anaesthetic, isoflurane will be recruited in this study. The medical and surgical care plans for participants remain as usual in this study with an exception being two additional blood samples of about two-teaspoonful in volume will be collected from an in-placed catheters in vein and aorta.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Two additional blood samples will be taken from in-situ catheters during heart surgery.

SUMMARY:
In the last few years, anaesthetic agents, Isoflurane used in heart surgery have shown some benefits to reduce the risk of heart muscle damage. Many research studies have been conducted to reveal the benefit relationship between Isoflurane and the risk of heart muscle injury during heart surgery. However, there is a knowledge gap regarding the optimal level of Isoflurane concentration to confer the benefit of heart muscle-protective properties. Therefore, this study is conducted to answer that question by measuring the Isoflurane concentration in the blood vessels. It also assesses whether Isoflurane concentration in the blood is correlated to the oxygenator exhaust level of Isoflurane in the heart-lung machine.

DETAILED DESCRIPTION:
All patients who scheduled for an elective heart surgery in Royal Infirmary of Edinburgh using a heart-lung machine and the administration of ether-like anaesthetic, isoflurane will be recruited in this study. This is a pilot study to determine the concentration of isoflurane in heart muscle. Isaac and Michael (2005), Hill (1998), Julious (2005) have conducted survey/research to conclude that 30 sample sizes are adequate for a pilot study. Thus, investigators aim to recruit at least 30 sample sizes to allow data (standard deviation, mean etc.) used in sample size estimation for future studies.

The medical and surgical care plans for participants remain as usual in this study. In a normal practise, surgeons will insert a catheter into the blood vessels coming from the heart to deliver solution to stop the contraction of heart for heart procedure. At this moment, two blood samples of about two-teaspoonful in volume will be collected from the in-placed catheters in vein and aorta. Then, the blood samples will be sent to lab to measure the concentration of isoflurane in vein and aorta. Also, the reading of exhausted isoflurane gas on heart-lung machine are routinely monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for elective cardiac surgery requiring cardiopulmonary bypass.
* Anaesthetised using isoflurane as part of a balanced anaesthetic technique during heart-lung machine
* Patient has consented to participate
* Cardioplegia technique involves insertion of a coronary sinus catheter.

Exclusion Criteria:

* Emergency surgery or patient with malignancy
* Heart surgery undertaken without heart-lung machine
* Age younger than 18 years
* Unable or unwilling to provide informed consent
* Cardiac surgery that does not require cardiopulmonary bypass
* Anaesthetised using an total intravenous-based technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who scheduled for an elective heart surgery in Royal Infirmary of Edinburgh using a heart-lung machine and the administration of ether-like anaesthetic, isoflurane will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Levels of Isoflurane in coronary sinus blood | 1 week after blood samples taken

SECONDARY OUTCOMES:
Isoflurane level in oxygenator exhaust levels on heart-lung machine | Immediately after the heart surgery is over

CONTACTS AND LOCATIONS:
Overall Officials: R Peter Alston, MB ChB, Principal Investigator — NHS Lothian
Locations (1):
- Department of Anaesthesia and Critical Care, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yau JM, Alexander JH, Hafley G, Mahaffey KW, Mack MJ, Kouchoukos N, Goyal A, Peterson ED, Gibson CM, Califf RM, Harrington RA, Ferguson TB; PREVENT IV Investigators. Impact of perioperative myocardial infarction on angiographic and clinical outcomes following coronary artery bypass grafting (from PRoject of Ex-vivo Vein graft ENgineering via Transfection [PREVENT] IV). Am J Cardiol. 2008 Sep 1;102(5):546-51. doi: 10.1016/j.amjcard.2008.04.069. Epub 2008 Jul 2. PMID 18721510
- [Background] BIGELOW WG, LINDSAY WK, GREENWOOD WF. Hypothermia; its possible role in cardiac surgery: an investigation of factors governing survival in dogs at low body temperatures. Ann Surg. 1950 Nov;132(5):849-66. doi: 10.1097/00000658-195011000-00001. No abstract available. PMID 14771796
- [Background] Yoshimi I. Cardiac preconditioning by anesthetic agents: roles of volatile anesthetics and opioids in cardioprotection. Yonago Acta Medica 2007; 50: 45-55.
- [Background] Hausenloy DJ, Boston-Griffiths E, Yellon DM. Cardioprotection during cardiac surgery. Cardiovasc Res. 2012 May 1;94(2):253-65. doi: 10.1093/cvr/cvs131. Epub 2012 Mar 22. PMID 22440888
- [Background] R. Peter Alston, Paul Myles, Marco Ranucci. Oxford Textbook of Cardiothoracic Anaesthesia. Oxford University Press 2015. Chapter 15 Myocardial protection during cardiac surgery. 157-65.
- [Background] Pramood CK, Reena S, Gajraj SS. Ischemic and anesthetic preconditioning of the heart: an insight into the concepts and mechanisms. Journal Indian Academy of Clinical Medicine; 2005; 6(1): 45-7
- [Background] Symons JA, Myles PS. Myocardial protection with volatile anaesthetic agents during coronary artery bypass surgery: a meta-analysis. Br J Anaesth. 2006 Aug;97(2):127-36. doi: 10.1093/bja/ael149. Epub 2006 Jun 21. PMID 16793778
- [Background] Fabien Picard, Francis Depret, Sergio ZC, Steven Hollenberg. Effect of anesthesia level on murine cardiac function. F1000 Research 2014; 3: 165-72
- [Background] Chiu-Fen Y, Michael Yu-Chih C, Tsung-I C, Ching-Feng Cheng. Dose-dependent effects of isoflurane on cardiovascular function in rats. Tzu Chi Medical Journal 2014; 26 (3): 119-22